CLINICAL TRIAL: NCT02146326
Title: The Impact of Burnout on Patient-Centered Care: A Comparative Effectiveness Trial in Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Four County Counseling Center (Unknown); Places for People (Unknown); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Michelle Salyers, Professor, Department of Psychology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IH-1304-6597
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Burnout; Quality of Care
MeSH Terms: conditions — Burnout, Psychological | interventions — Motivational Interviewing; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Motivational Interviewing-Mental Health Staff (Active Comparator)
  Interventions: Behavioral: Motivational Interviewing (MI)
- BREATHE-Mental Health Staff (Active Comparator)
  Interventions: Behavioral: Burnout Reduction: Enhanced Awareness, Tools, Handouts, and Education (BREATHE)
- Motivational Interviewing-Clients (Active Comparator)
  Interventions: Behavioral: Motivational Interviewing (MI)
- BREATHE-Clients (Active Comparator)
  Interventions: Behavioral: Burnout Reduction: Enhanced Awareness, Tools, Handouts, and Education (BREATHE)

INTERVENTIONS:
Behavioral: Motivational Interviewing (MI) — MI is a common counseling technique. It was offered as an 8-9 hour workshop across 3 sessions to mental health agency staff who were randomly assigned to MI. Each session occurred approximately one month apart.
  Arms: Motivational Interviewing-Clients; Motivational Interviewing-Mental Health Staff
Behavioral: Burnout Reduction: Enhanced Awareness, Tools, Handouts, and Education (BREATHE) — BREATHE is a program developed to attempt to improve or prevent the symptoms of burnout. It was offered as an 8-9 hour workshop across 3 sessions to mental health agency staff who were randomly assigned to BREATHE. Each session occurred approximately one month apart.
  Arms: BREATHE-Clients; BREATHE-Mental Health Staff

SUMMARY:
Healthcare providers play an important role in helping patients be actively involved in treatment and recover from mental illness. But mental health clinicians, like other healthcare providers, are at risk for experiencing burnout-feeling emotionally drained from their work, having cynical thoughts toward patients and others, and feeling little accomplishment in their work. Burnout can lead to problems for the clinician including poor overall health, depression, and lower job satisfaction. Burnout also can impact how clinicians perform on the job; for example, people with high levels of burnout take more time off, show lower commitment to their job, and are more likely to quit or be fired. There is some evidence that burnout can affect the quality of care for patients, but very little rigorous research has tested this assumption. The purpose of our study is threefold. First, we will investigate how patients perceive burnout in clinicians and whether (and/or how) burnout impacts the care they receive. Next, we will test an intervention to reduce clinician burnout called Burnout Reduction: Enhanced Awareness, Tools, Handouts, and Education (BREATHE). BREATHE brings together tools that mental health clinicians are already familiar with, including relaxation and mindfulness exercises, setting boundaries, using social supports, and changing negative thought patterns and replacing them with more helpful ways of thinking. We have found this intervention effective in reducing burnout in other organizations, but have yet to study whether it also can improve patient outcomes. Clinicians (approximately 200) who participate will receive either the BREATHE intervention or training in motivational interviewing, which could also improve patient involvement in treatment and patient outcomes, but is unlikely to significantly reduce clinician burnout. We will also recruit up to 600 adult patients served by participating clinicians. We will survey clinicians and interview patients over a 12-month period after the intervention to determine how the intervention impacts clinician burnout and patient perceptions of care (relationship with the clinician, degree of autonomy in decision making), patient involvement in care, and outcomes (confidence in managing mental health, symptoms, functioning, and hope). Finally, this study will use a statistical procedure called Structural Equation Modeling to test a theoretical model of the relationship between burnout and patient outcomes. Findings from this study will show whether reducing clinician burnout can improve patient outcomes and the quality of care that patients receive. Our intervention will have the potential to be easily implemented in a variety of settings where burnout is a problem. Knowing how clinician burnout impacts patient outcomes, and whether improving burnout can improve patient care, can help improve the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* A staff member with client contact at either Four County Counseling or Places for People.
* Randomly chosen client from the participating staff lists. Must be 18 years old or older.

Exclusion Criteria:

* Clients younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 679 (Actual)
Dates: Start 2013-12; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle P Salyers, PhD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Four County Counseling Center, Logansport, Indiana
  - Places for People, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Staff and clients were recruited from 2 community mental health centers. Up to 5 clients for each participating staff with adult caseloads were recruited. Enrollment occurred over 3 waves of recruitment at 2 sites between 2/24/2014 and 3/18/2016. Totals of 206 staff and 473 clients completed informed consent to participate.
Pre-assignment Details: Mental Health Care Staff:
  206 completed informed consent: 14 were not randomized (12 did not complete the baseline survey, 1 withdrew, 1 resigned), 192 staff were randomized
  Mental Health Clients:
  473 clients completed informed consent: 4 were not linked to randomized staff (3 screen failures, 1 linked to staff not randomized),
Groups:
- BREATHE-Mental Health Care Staff: Mental Health Care Staff randomized to the Burnout Reduction: Enhanced Awareness, Tools, Handouts, and Education (BREATHE) intervention:
  Staff were invited to attend an 8-9 hour BREATHE workshop delivered in 3 sessions, each about one month apart. Staff were asked to complete online surveys at the following time points: Baseline, 3 months, 6 months, and 12 months.
- Motivational Interviewing-Mental Health Care Staff: Mental Health Care Staff randomized to the Motivational Interviewing (MI) intervention:
  Staff were invited to attend an 8-9 hour MI workshop delivered in 3 sessions, each about one month apart. Staff were asked to complete online surveys at the following time points: Baseline, 3 months, 6 months, and 12 months.
- BREATHE-Clients: Clients linked to staff randomized to the BREATHE intervention:
  Clients were invited to be interviewed at the following time points: Baseline, 6 months, and 12 months.
- Motivational Interviewing-Clients: Clients linked to staff randomized to the MI intervention:
  Clients were invited to be interviewed at the following time points: Baseline, 6 months, and 12 months.
Period: Overall Study
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Started | 89 | 103 | 211 | 258
Baseline | 89 | 103 | 211 | 258
3 Months | 71 | 83 | 0 | 0
6 Months | 71 | 71 | 186 | 235
12 Months | 61 | 66 | 168 | 210
Completed | 61 | 66 | 168 | 210
Not Completed | 28 | 37 | 43 | 48
Not completed — Lost to Follow-up | 3 | 3 | 11 | 19
Not completed — Withdrawal by Subject | 2 | 1 | 15 | 11
Not completed — Separated from mental health center | 23 | 33 | 0 | 0
Not completed — Incarcerated | 0 | 0 | 3 | 8
Not completed — Death | 0 | 0 | 4 | 4
Not completed — Unable to complete interview | 0 | 0 | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- BREATHE-Mental Health Care Staff: Mental Health Care Staff randomized to the BREATHE intervention: Staff were invited to attend an 8-9 hour BREATHE workshop delivered in 3 sessions, each about one month apart. Staff were asked to complete online surveys at the following time points: Baseline, 3 months, 6 months, and 12 months.
- Motivational Interviewing-Mental Health Care Staff: Mental Health Care Staff randomized to the MI intervention: Staff were invited to attend an 8-9 hour MI workshop delivered in 3 sessions, each about one month apart. Staff were asked to complete online surveys at the following time points: Baseline, 3 months, 6 months, and 12 months.
- Total: Total of all reporting groups
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients | Total
Number analyzed (Participants) | 89 | 103 | 211 | 258 | 661
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of staff population. Population: Age of client population reported separately.
  years
    number analyzed (Participants) | 89 | 103 | 0 | 0 | 192
    (all) | 41.3 (12.5) | 39.5 (12.0) |  |  | 40.3 (12.2)
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of client population. Population: Age of staff population reported separately.
  years
    number analyzed (Participants) | 0 | 0 | 211 | 258 | 469
    (all) |  |  | 45.2 (13.6) | 45.2 (12.7) | 45.2 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 89 | 104 | 138 | 395
  Male | 25 | 14 | 107 | 120 | 266
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 13 | 6 | 84 | 118 | 221
  White | 71 | 91 | 115 | 129 | 406
  Other | 4 | 6 | 12 | 9 | 31
  Missing/Unknown | 1 | 0 | 0 | 0 | 1
Education (Staff) [Count of Participants; unit: Participants] — Highest level of education (staff) Population: Education was analyzed in relation to bachelors degree for staff only. Education for clients was analyzed in relation to High School/GED completion and is reported separately.
  Participants
    Bachelors degree or above: number analyzed (Participants) | 89 | 103 | 0 | 0 | 192
    Bachelors degree or above | 69 | 88 |  |  | 157
    Less than bachelors degree: number analyzed (Participants) | 89 | 103 | 0 | 0 | 192
    Less than bachelors degree | 20 | 14 |  |  | 34
    Missing/Unknown: number analyzed (Participants) | 89 | 103 | 0 | 0 | 192
    Missing/Unknown | 0 | 1 |  |  | 1
Education (Clients) [Count of Participants; unit: Participants] — Highest grade of school completed (clients) Population: Education was analyzed in relation to completion of high school/GED for the client population only. Education for staff was analyzed in relation to bachelors degree or above and is reported separately.
  Participants
    Completed at least high school/GED: number analyzed (Participants) | 0 | 0 | 211 | 258 | 469
    Completed at least high school/GED |  |  | 150 | 178 | 328
    Less than high school/GED: number analyzed (Participants) | 0 | 0 | 211 | 258 | 469
    Less than high school/GED |  |  | 61 | 80 | 141
Years in position (Staff) [Mean (Standard Deviation); unit: years] — Staff answered the question: "How long have you been in your current position? (in years)" Population: This only applies to the staff population. One participant did not answer the question.
  years
    number analyzed (Participants) | 89 | 102 | 0 | 0 | 191
    (all) | 3.5 (4.7) | 3.1 (4.7) |  |  | 3.3 (4.7)
Years at agency (Staff) [Mean (Standard Deviation); unit: years] — Staff were asked: How long have you been at Four County/Places for People? (in years) Population: This only applies to the staff population. One participant did not answser the question.
  years
    number analyzed (Participants) | 89 | 102 | 0 | 0 | 191
    (all) | 4.8 (5.7) | 5.3 (6.7) |  |  | 5.0 (6.3)
Percentage of interactions with adult clients (Staff) [Count of Participants; unit: Participants] — Staff were asked what percentage of client interactions are with adult clients (aged 18 or older). The data include those who reported at least 1%. Population: This only applies to staff participants. One participant did not answer the question.
  Participants
    number analyzed (Participants) | 89 | 102 | 0 | 0 | 191
    (all) | 80 | 94 |  |  | 174
Years in field (Staff) [Mean (Standard Deviation); unit: years] — Staff were asked how long they had been working in the mental health field (in years). Population: This only applies to the staff population. Two participants did not answer the question.
  years
    number analyzed (Participants) | 89 | 101 | 0 | 0 | 190
    (all) | 9.4 (9.2) | 8.4 (8.8) |  |  | 8.9 (9.0)
Hours of burnout training in past year (Staff) [Mean (Standard Deviation); unit: hours] — Staff were asked how much training in burnout prevention/reduction they had received in the past year. Population: This only applies to the staff population. Four participants (two from each condition) did not answer this question.
  hours
    number analyzed (Participants) | 87 | 101 | 0 | 0 | 188
    (all) | 0.7 (3.4) | 0.8 (2.4) |  |  | 0.8 (2.9)
Hours of motivational interviewing training in past year (Staff) [Mean (Standard Deviation); unit: hours] — Staff were asked how much training in motivational interviewing they had received in the past year. Population: This only applies to the staff population. Three participants (1 assigned to BREATHE and 2 assigned to MI) did not answer the question.
  hours
    number analyzed (Participants) | 88 | 101 | 0 | 0 | 189
    (all) | 3.1 (8.2) | 1.9 (4.5) |  |  | 2.5 (6.5)
Official number of work hours (Staff) [Mean (Standard Deviation); unit: hours] — Staff were asked how many official hours they are scheduled to work in a typical work week. Population: This only applies to the staff population. One participant did not answer the question.
  hours
    number analyzed (Participants) | 89 | 102 | 0 | 0 | 191
    (all) | 39.1 (4.6) | 38.5 (5.4) |  |  | 38.8 (5.0)
Actual number of work hours (Staff) [Mean (Standard Deviation); unit: hours] — Staff were asked how many hours they actually work in a typical work week. One participant did not answer the question. Population: This only applies to the staff population.
  hours
    number analyzed (Participants) | 89 | 102 | 0 | 0 | 191
    (all) | 41.6 (6.4) | 41.6 (7.0) |  |  | 41.6 (6.7)
Employment (Clients) [Count of Participants; unit: Participants] — Clients were asked if they were currently employed. Response choices were paid employment, casual work (i.e., babysitting, side jobs, etc.), student, unemployed and looking for work, unemployed and not looking for work, other, refused. Population: This measure only applies to the client population.
  Participants
    number analyzed (Participants) | 0 | 0 | 211 | 258 | 469
    Paid employment |  |  | 26 | 36 | 62
    Other |  |  | 185 | 222 | 407
Housing (Clients) [Count of Participants; unit: Participants] — Clients were asked what type of housing they currently live in. Housing codes included: homeless-on streets or in shelter, staying with friends or family temporarily, structured congregate living (e.g., nursing home, group home, residential facilities), semi-independing living (staff member lives on site, or foster family care), living with family (not spouse), own apartment or house (with spouse, living as married, with friends), own apartment or house-alone (includes boarding homes, hotels) Population: This only applies to the client population.
  Participants
    number analyzed (Participants) | 0 | 0 | 211 | 258 | 469
    Independent living |  |  | 143 | 161 | 304
    Other |  |  | 68 | 97 | 165
Required to attend treatment (Clients) [Count of Participants; unit: Participants] — Clients were asked if they were required to attend treatment at the agency due to involuntary commitment, court order, or other legal requirement. Population: This only applies to the client population.
  Participants
    number analyzed (Participants) | 0 | 0 | 211 | 258 | 469
    Yes, required to attend treatment | 0 | 0 | 30 | 50 | 80
    No, not required or unknown/refused | 0 | 0 | 181 | 208 | 389
Wants to attend treatment (Clients) [Count of Participants; unit: Participants] — Clients were asked if they want to attend treatment. Population: This only applies to the client population.
  Participants
    number analyzed (Participants) | 0 | 0 | 211 | 258 | 469
    Yes, want to attend treatment | 0 | 0 | 197 | 236 | 433
    No, does not want or unknown/refused | 0 | 0 | 14 | 22 | 36
Primary Diagnosis Category (Clients) [Count of Participants; unit: Participants] — Diagnosis information from client medical records were reviewed to determine the most common primary mental health diagnosis category. Population: This only applies to the client population.
  Participants
    Anxiety Disorder: number analyzed (Participants) | 0 | 0 | 211 | 258 | 469
    Anxiety Disorder |  |  | 19 | 12 | 31
    Bipolar Disorder: number analyzed (Participants) | 0 | 0 | 211 | 258 | 469
    Bipolar Disorder |  |  | 35 | 45 | 80
    Major Depression: number analyzed (Participants) | 0 | 0 | 211 | 258 | 469
    Major Depression |  |  | 55 | 53 | 108
    Other: number analyzed (Participants) | 0 | 0 | 211 | 258 | 469
    Other |  |  | 8 | 12 | 20
    Schizophrenia: number analyzed (Participants) | 0 | 0 | 211 | 258 | 469
    Schizophrenia |  |  | 86 | 127 | 213
    Missing/Unknown: number analyzed (Participants) | 0 | 0 | 211 | 258 | 469
    Missing/Unknown |  |  | 8 | 9 | 17
Substance Use (Clients) [Count of Participants; unit: Participants] — Diagnosis information from client medical record data were reviewed for the presence of any substance use diagnoses (excluding tobacco/nicotine only). Population: This only applies to the client population.
  Participants
    Substance Use Not Present: number analyzed (Participants) | 0 | 0 | 211 | 258 | 469
    Substance Use Not Present |  |  | 142 | 169 | 311
    Substance Use Present: number analyzed (Participants) | 0 | 0 | 211 | 258 | 469
    Substance Use Present |  |  | 60 | 80 | 140
    Missing/Unknown: number analyzed (Participants) | 0 | 0 | 211 | 258 | 469
    Missing/Unknown |  |  | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Maslach Burnout Inventory (MBI): Emotional Exhaustion
Description: Burnout was assessed with the Maslach Burnout Inventory (MBI), a widely-used measure of three components of burnout: emotional exhaustion, depersonalization, and personal accomplishment. The survey contains 22 statements of job-related feelings and staff were asked to read each statement and decide if they ever felt that way about their job. The item scores were averaged. Scale: 0 (Never), 1 (A few times a year or less), 2 (Once a month or less), 3 (A few times a month), 4 (Once a week), 5 (A few times a week), 6 (Every Day).
  Maslach C, Jackson, S. E., Leiter, M. P. Maslach Burnout Inventory Manual. 3 ed. Palo Alto, California: Consulting Psychologists Press; 1996.
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: The number analyzed at each time point differs from the overall number enrolled due to participant drop out and/or missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 89 | 102 | 0 | 0
  Baseline | 2.3 (1.3) | 2.7 (1.3) |  |
  3 months: number analyzed (Participants) | 72 | 83 | 0 | 0
  3 months | 2.3 (1.2) | 2.7 (1.4) |  |
  6 months: number analyzed (Participants) | 71 | 71 | 0 | 0
  6 months | 2.5 (1.4) | 2.6 (1.3) |  |
  12 months: number analyzed (Participants) | 61 | 66 | 0 | 0
  12 months | 2.4 (1.2) | 2.5 (1.3) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; Mixed effects regression analysis was used to examine the BREATHE intervention effect on clinician burnout and patient processes, engagement, and outcomes as compared to MI after the intervention by adjusting for the baseline scores and the implementation site; Test type: Superiority; p = 0.80, Mixed Models Analysis

2. Primary Outcome: Maslach Burnout Inventory (MBI): Depersonalization
Description: Burnout was assessed with the Maslach Burnout Inventory (MBI), a widely-used measure of three components of burnout: emotional exhaustion, depersonalization, and personal accomplishment. The survey contains 22 statements of job-related feelings and staff were ased to read each statement and decide if they ever felt that way about their job. The item scores were averaged. Scale: 0 (Never), 1 (A few times a year or less), 2 (Once a month or less), 3 (A few times a month), 4 (Once a week), 5 (A few times a week), 6 (Every Day).
  Maslach C, Jackson, S. E., Leiter, M. P. Maslach Burnout Inventory Manual. 3 ed. Palo Alto, California: Consulting Psychologists Press; 1996.
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: The number analyzed at each time point differs from the overall number due to participant drop out and/or missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 89 | 102 | 0 | 0
  Baseline | 1.3 (0.9) | 1.5 (1.1) |  |
  3 months: number analyzed (Participants) | 72 | 83 | 0 | 0
  3 months | 1.2 (0.8) | 1.4 (1.0) |  |
  6 months: number analyzed (Participants) | 71 | 71 | 0 | 0
  6 months | 1.3 (0.9) | 1.5 (1.2) |  |
  12 months: number analyzed (Participants) | 60 | 66 | 0 | 0
  12 months | 1.3 (1.1) | 1.3 (0.9) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.80, Mixed Models Analysis

3. Primary Outcome: Maslach Burnout Inventory (MBI): Personal Accomplishment
Description: as for outcome 2
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 89 | 102 | 0 | 0
  Baseline | 4.9 (0.8) | 4.9 (0.7) |  |
  3 months: number analyzed (Participants) | 72 | 83 | 0 | 0
  3 months | 4.9 (0.7) | 4.9 (0.7) |  |
  6 months: number analyzed (Participants) | 71 | 71 | 0 | 0
  6 months | 4.9 (0.9) | 4.9 (0.7) |  |
  12 months: number analyzed (Participants) | 60 | 66 | 0 | 0
  12 months | 4.8 (0.8) | 4.8 (0.8) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.54, Mixed Models Analysis

4. Secondary Outcome: Job Satisfaction
Description: Job satisfaction was assessed with one item from the Job Diagnostics Survey: Overall, I am satisfied with my job. Scale: 1 (Strongly Disagree) to 7 (Strongly Agree)
  Hackman JR, Oldham GR. The Job Diagnostic Survey: An Instrument for the Diagnosis of Jobs and the Evaluation of Job Redesign Projects. 1974.
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 82 | 94 | 0 | 0
  Baseline | 5.7 (1.4) | 5.2 (1.6) |  |
  3 months: number analyzed (Participants) | 61 | 67 | 0 | 0
  3 months | 5.4 (1.6) | 5.1 (1.5) |  |
  6 months: number analyzed (Participants) | 61 | 59 | 0 | 0
  6 months | 5.3 (1.7) | 4.9 (1.7) |  |
  12 months: number analyzed (Participants) | 59 | 58 | 0 | 0
  12 months | 5.6 (1.4) | 5.2 (1.5) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.94, Mixed Models Analysis

5. Secondary Outcome: Turnover Intentions-Considered Leaving
Description: This is the first of two questions in which staff were asked about turnover intentions. Staff were asked, "How often have you seriously considered leaving your job in the past six months?" Scale: 1 (Never), 2 (Once every few months), 3 (Once a month), 4 (several times a month), 5 (Once a week), 6 (Several times a week)
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 89 | 102 | 0 | 0
  Baseline | 2.0 (1.2) | 2.6 (1.7) |  |
  3 months: number analyzed (Participants) | 71 | 83 | 0 | 0
  3 months | 2.4 (1.4) | 2.6 (1.6) |  |
  6 months: number analyzed (Participants) | 70 | 71 | 0 | 0
  6 months | 2.5 (1.7) | 2.8 (1.8) |  |
  12 months: number analyzed (Participants) | 61 | 66 | 0 | 0
  12 months | 2.6 (1.5) | 2.7 (1.6) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.96, Mixed Models Analysis

6. Secondary Outcome: Turnover Intentions-Likely to Leave
Description: This is the second of two questions in which staff were asked about turnover intentions. Staff were asked, "How likely are you to leave your job in the next six months?" Scale: 1 (Not likely at all), 2 (Not very likely), 3 (Somewhat likely), 4 (Very likely)
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 89 | 102 | 0 | 0
  Baseline | 1.6 (0.8) | 1.9 (1.0) |  |
  3 months: number analyzed (Participants) | 72 | 83 | 0 | 0
  3 months | 1.8 (1.0) | 2.0 (1.0) |  |
  6 months: number analyzed (Participants) | 70 | 71 | 0 | 0
  6 months | 1.9 (1.0) | 2.2 (1.0) |  |
  12 months: number analyzed (Participants) | 60 | 66 | 0 | 0
  12 months | 1.8 (0.9) | 2.1 (1.1) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.17, Mixed Models Analysis

7. Secondary Outcome: Work Interference With Home Life
Description: Work-Life Balance was assessed with a six-item measure adapted from an 18-item measure developed by Carlson et al. The measure assesses three types (time-, strain-, and behavior-based) and two directions (work conflict with family and family conflict with work) of balance. The outcome described here is work conflict with family. The measure consists of a series of statements regarding one's work and family situation, to which participants are asked to indicate their level of agreement or disagreement on a 5-point Likert-type scale: 1 (Strongly disagree) to 5 (Strongly agree). The item scores were averaged.
  Carlson DS, Kacmar KM, Williams LJ. Construction and initial validation of a multidimensional measure of work-family conflict. Journal of Vocational Behavior. 2000;56(2):249-276.
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Motivational Interviewing-Mental Health Care Staff: Mental Health Care Staff randomized to the MI intervention Staff were invited to attend an 8-9 hour MI workshop delivered in 3 sessions, each about one month apart. Staff were asked to complete online surveys at the following time points: Baseline, 3 months, 6 months, and 12 months.
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 89 | 102 | 0 | 0
  Baseline | 2.7 (0.9) | 2.9 (1.0) |  |
  3 months: number analyzed (Participants) | 71 | 83 | 0 | 0
  3 months | 2.7 (0.9) | 2.9 (1.1) |  |
  6 months: number analyzed (Participants) | 71 | 70 | 0 | 0
  6 months | 2.7 (1.0) | 2.9 (1.0) |  |
  12 months: number analyzed (Participants) | 61 | 65 | 0 | 0
  12 months | 2.7 (0.8) | 2.9 (1.0) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.47, Mixed Models Analysis

8. Secondary Outcome: Home Life Interference With Work
Description: Work-Life Balance was assessed with a six-item measure adapted from an 18-item measure developed by Carlson et al. The measure assesses three types (time-, strain-, and behavior-based) and two directions (work conflict with family and family conflict with work) of balance. The outcome described here is family conflict with work. The measure consists of a series of statements regarding one's work and family situation, to which participants are asked to indicate their level of agreement or disagreement on a 5-point Likert-type scale: 1 (Strongly disagree) to 5 (Strongly agree). The item scores were averaged.
  Carlson DS, Kacmar KM, Williams LJ. Construction and initial validation of a multidimensional measure of work-family conflict. Journal of Vocational Behavior. 2000;56(2):249-276.
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 89 | 102 | 0 | 0
  Baseline | 1.9 (0.7) | 1.9 (0.7) |  |
  3 months: number analyzed (Participants) | 71 | 83 | 0 | 0
  3 months | 1.8 (0.7) | 1.9 (0.7) |  |
  6 months: number analyzed (Participants) | 71 | 70 | 0 | 0
  6 months | 1.9 (0.8) | 1.8 (0.7) |  |
  12 months: number analyzed (Participants) | 61 | 65 | 0 | 0
  12 months | 1.9 (0.7) | 1.8 (0.7) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.60, Mixed Models Analysis

9. Secondary Outcome: Emotional Labor Scale: Surface Acting
Description: The Emotional Labor Scale includes 14 questions regarding the relationship between emotions and interactions with clients. Surface Acting is a subset of these questions (e.g., I put on an act in order to deal with clients in an appropriate way). The item scores were averaged. Scale: 1 (strongly disagree) to 5 (strongly agree)
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 89 | 102 | 0 | 0
  Baseline | 2.1 (0.8) | 2.2 (0.8) |  |
  3 months: number analyzed (Participants) | 72 | 83 | 0 | 0
  3 months | 2.2 (0.8) | 2.3 (0.9) |  |
  6 months: number analyzed (Participants) | 71 | 71 | 0 | 0
  6 months | 2.1 (0.9) | 2.2 (1.0) |  |
  12 months: number analyzed (Participants) | 60 | 66 | 0 | 0
  12 months | 2.2 (0.9) | 2.1 (0.9) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.37, Mixed Models Analysis

10. Secondary Outcome: Emotional Labor Scale: Deep Acting
Description: The Emotional Labor Scale includes 14 questions regarding the relationship between emotions and interactions with clients. Deep Acting is a subset of these questions (e.g., I try to actually experience the emotions that I must show to clients). The item scores were averaged. Scale: 1 (strongly disagree) to 5 (strongly agree)
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 89 | 102 | 0 | 0
  Baseline | 3.4 (0.9) | 3.2 (0.9) |  |
  3 months: number analyzed (Participants) | 72 | 83 | 0 | 0
  3 months | 3.4 (0.7) | 3.1 (1.0) |  |
  6 months: number analyzed (Participants) | 71 | 71 | 0 | 0
  6 months | 3.1 (0.9) | 3.2 (1.0) |  |
  12 months: number analyzed (Participants) | 60 | 66 | 0 | 0
  12 months | 3.2 (0.8) | 3.0 (1.0) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.83, Mixed Models Analysis

11. Secondary Outcome: Emotional Labor Scale: Genuine Emotions
Description: The Emotional Labor Scale includes 14 questions regarding the relationship between emotions and interactions with clients. Genuine Emotions is a subset of these questions (e.g., The emotions that I express to clients are genuine). The item scores were averaged. Scale: 1 (strongly disagree) to 5 (strongly agree)
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 89 | 102 | 0 | 0
  Baseline | 4.0 (0.8) | 4.0 (0.6) |  |
  3 months: number analyzed (Participants) | 72 | 82 | 0 | 0
  3 months | 4.1 (0.8) | 4.0 (0.7) |  |
  6 months: number analyzed (Participants) | 71 | 71 | 0 | 0
  6 months | 3.9 (0.7) | 4.0 (0.8) |  |
  12 months: number analyzed (Participants) | 60 | 66 | 0 | 0
  12 months | 4.0 (0.7) | 4.1 (0.7) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.64, Mixed Models Analysis

12. Secondary Outcome: Importance: Reduce Work-Related Stress
Description: Staff were asked, "How important is it for you to reduce your work-related stress right now?" This single item score was averaged. Scale: 1 (not at all important) to 10 (extremely important)
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 89 | 102 | 0 | 0
  Baseline | 6.5 (3.0) | 6.4 (2.8) |  |
  3 months: number analyzed (Participants) | 70 | 83 | 0 | 0
  3 months | 6.4 (2.9) | 7.3 (2.6) |  |
  6 months: number analyzed (Participants) | 71 | 71 | 0 | 0
  6 months | 6.5 (3.0) | 7.5 (2.6) |  |
  12 months: number analyzed (Participants) | 61 | 66 | 0 | 0
  12 months | 6.6 (2.8) | 6.6 (3.0) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.37, Mixed Models Analysis

13. Secondary Outcome: Confidence: Reduce Work-Related Stress
Description: Staff were asked, "How confident are you that you can reduce your work-related stress in your life?" Scale: 1 (not at all confident) to 10 (extremely confident)
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 89 | 102 | 0 | 0
  Baseline | 7.0 (2.3) | 6.0 (2.6) |  |
  3 months: number analyzed (Participants) | 72 | 83 | 0 | 0
  3 months | 6.5 (2.6) | 6.3 (2.5) |  |
  6 months: number analyzed (Participants) | 71 | 71 | 0 | 0
  6 months | 6.6 (2.5) | 5.7 (2.5) |  |
  12 months: number analyzed (Participants) | 61 | 66 | 0 | 0
  12 months | 6.5 (2.8) | 5.5 (2.6) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.13, Mixed Models Analysis

14. Secondary Outcome: Importance: Client Interaction
Description: Staff were asked, "How important is it for you to consistently interact with consumers/clients in a relaxed, non-judgmental way?" Scale: 1 (not at all important) to 10 (extremely important)
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 89 | 102 | 0 | 0
  Baseline | 9.4 (1.0) | 9.5 (1.2) |  |
  3 months: number analyzed (Participants) | 72 | 83 | 0 | 0
  3 months | 9.5 (0.9) | 9.3 (1.3) |  |
  6 months: number analyzed (Participants) | 71 | 69 | 0 | 0
  6 months | 9.3 (1.2) | 9.2 (1.8) |  |
  12 months: number analyzed (Participants) | 59 | 65 | 0 | 0
  12 months | 9.3 (1.2) | 9.3 (1.7) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.93, Mixed Models Analysis

15. Secondary Outcome: Confidence: Client Interaction
Description: Staff were asked, "How confident are you that you can consistently interact with consumers/clients in a relaxed, non-judgmental way?" Scale: 1 (not at all confident) to 10 (extremely confident)
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 89 | 101 | 0 | 0
  Baseline | 8.5 (1.5) | 8.3 (1.7) |  |
  3 months: number analyzed (Participants) | 72 | 83 | 0 | 0
  3 months | 8.5 (1.5) | 8.1 (1.7) |  |
  6 months: number analyzed (Participants) | 71 | 70 | 0 | 0
  6 months | 8.5 (1.4) | 8.1 (1.7) |  |
  12 months: number analyzed (Participants) | 59 | 66 | 0 | 0
  12 months | 8.8 (1.4) | 8.2 (1.9) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.11, Mixed Models Analysis

16. Secondary Outcome: Quality of Care: Person Centered Care
Description: Perceived Quality of Care was assessed with a 31 item scale developed with one of the mental health agencies as part of this project. Person Centered Care was measured with a subset of questions from this scale (e.g., I felt like I was able to really show compassion to a client.). The item scores were averaged. Scale: 0 (never) to 5 (always)
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 86 | 99 | 0 | 0
  Baseline | 3.7 (0.8) | 3.6 (0.6) |  |
  3 months: number analyzed (Participants) | 71 | 82 | 0 | 0
  3 months | 3.8 (0.6) | 3.7 (0.6) |  |
  6 months: number analyzed (Participants) | 71 | 70 | 0 | 0
  6 months | 3.8 (0.6) | 3.8 (0.6) |  |
  12 months: number analyzed (Participants) | 58 | 65 | 0 | 0
  12 months | 3.8 (0.6) | 3.8 (0.6) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.21, Mixed Models Analysis

17. Secondary Outcome: Quality of Care: Discordant Care
Description: Perceived Quality of Care was assessed with a 31 item scale developed with one of the mental health agencies as part of this project. Discordant Care was measured with a subset of questions from this scale (e.g., I had conflicts with clients.). The item scores were averaged. Scale: 0 (never) to 5 (always)
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 88 | 101 | 0 | 0
  Baseline | 3.8 (0.5) | 3.8 (0.5) |  |
  3 months: number analyzed (Participants) | 71 | 83 | 0 | 0
  3 months | 3.8 (0.5) | 3.8 (0.6) |  |
  6 months: number analyzed (Participants) | 70 | 71 | 0 | 0
  6 months | 3.9 (0.5) | 3.8 (0.7) |  |
  12 months: number analyzed (Participants) | 61 | 65 | 0 | 0
  12 months | 3.8 (0.6) | 3.9 (0.5) |  |

18. Secondary Outcome: Quality of Care-Total
Description: Perceived Quality of Care was assessed with a 31 item scale developed with one of the mental health agencies participating in this project and then refined to 22 items through data collected and analyzed in this study. Items were related to person or client centered care, work conscientiousness, errors, interactions with clients, and how stress affects client interactions or outcomes. The item scores were averaged. Scale: 0 (never) to 5 (always)
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Motivational Interviewing-Clients: Clients linked to staff randomized to the MI intervention Clients: were invited to be interviewed at the following time points: Baseline, 6 months, and 12 months.
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 87 | 100 | 0 | 0
  Baseline | 3.8 (0.5) | 3.7 (0.5) |  |
  3 months: number analyzed (Participants) | 71 | 83 | 0 | 0
  3 months | 3.8 (0.4) | 3.7 (0.5) |  |
  6 months: number analyzed (Participants) | 71 | 71 | 0 | 0
  6 months | 3.8 (0.5) | 3.8 (0.5) |  |
  12 months: number analyzed (Participants) | 61 | 65 | 0 | 0
  12 months | 3.8 (0.5) | 3.9 (0.4) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.17, Mixed Models Analysis

19. Secondary Outcome: Perceptions of Supervisory Support
Description: The 19 item Perceptions of Supervisory Support Scale was used to gather information on staff's experience of interactions with their supervisors (e.g., How often did you think supervision improved your relationship with your supervisor?). The item scores were averaged. Scale: 1 (never) to 6 (always)
Time Frame: Measured with staff at baseline, 3 months, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
units on a scale
  Baseline: number analyzed (Participants) | 87 | 100 | 0 | 0
  Baseline | 4.1 (1.1) | 3.9 (1.0) |  |
  3 months: number analyzed (Participants) | 71 | 83 | 0 | 0
  3 months | 4.0 (1.2) | 3.9 (1.0) |  |
  6 months: number analyzed (Participants) | 70 | 71 | 0 | 0
  6 months | 3.9 (1.2) | 3.8 (1.0) |  |
  12 months: number analyzed (Participants) | 61 | 65 | 0 | 0
  12 months | 4.0 (1.1) | 4.0 (1.2) |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; Test type: Superiority; p = 0.24, Mixed Models Analysis

20. Secondary Outcome: Staff Turnover
Description: Number of staff participants who separated from their respective agency before their anticipated study completion date. The mental health agencies provided separation dates, if applicable, for staff study participants.
Time Frame: Measured with staff at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 89 | 103 | 0 | 0
Participants
  Separated from Agency | 23 | 33 |  |
  Not Separated from Agency | 66 | 70 |  |
Statistical Analysis 1: Comparison: BREATHE-Mental Health Care Staff vs Motivational Interviewing-Mental Health Care Staff; Test type: Superiority; p = 0.35, Chi-squared

21. Secondary Outcome: Adult State Hope Scale
Description: Hope was assessed with clients using the 12-item Adult State Hope Scale (e.g., I can think of many ways to get the things in life that are most important to me.). The item scores were averaged. Scale: 1 (Definitely False) to 8 (Definitely True)
  Snyder CR, Sympson SC, Ybasco FC, Borders TF, Babyak MA, Higgins RL. Development and validation of the State Hope Scale. Journal of Personality and Social Psychology. 1996;70(2):321 - 335.
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline |  |  | 5.78 (1.3) | 5.78 (1.2)
  6 months: number analyzed (Participants) | 0 | 0 | 185 | 235
  6 months |  |  | 5.75 (1.3) | 5.85 (1.2)
  12 months: number analyzed (Participants) | 0 | 0 | 164 | 207
  12 months |  |  | 5.77 (1.3) | 5.85 (1.1)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; Mixed effects regression analysis was used to examine the BREATHE intervention effect on patient processes, engagement, and outcomes as compared to MI after the intervention by adjusting for the baseline scores and the implementation site; Test type: Superiority; p = 0.67, Mixed Models Analysis

22. Secondary Outcome: Medication Adherence Rating Scale (MARS) - Medication Adherence - 4-item
Description: Medication adherence (for clients who are prescribed medications for their mental health) was rated with a subset of 4 items from the MARS, a 10-item scale assessing attitudes toward medication (e.g., Do you ever forget to take your medication? Are you careless at times about taking your medicine?). The item scores were summed and averaged (range: 0-4). Scale: 0 (No) to 1 (Yes)
  Thompson K, Kulkarni J, Sergejew AA. Reliability and validity of a new Medication Adherence Rating Scale (MARS) for the psychoses. Schizophrenia Research. May 5 2000;42(3):241-247.
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: The number analyzed at each time point differs from the overall number enrolled due to participant drop out, clients reporting they are not prescribed medications for their mental health, and/or missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 125 | 154
  Baseline |  |  | 1.9 (1.0) | 2.0 (1.0)
  6 months: number analyzed (Participants) | 0 | 0 | 99 | 144
  6 months |  |  | 1.8 (1.0) | 2.0 (1.1)
  12 months: number analyzed (Participants) | 0 | 0 | 93 | 111
  12 months |  |  | 1.6 (0.9) | 1.9 (1.1)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.04, Mixed Models Analysis

23. Secondary Outcome: Medication Adherence Rating Scale (MARS) - Medication Attitudes - 10-item
Description: Medication attitudes (for clients who are prescribed medications for their mental health) was rated with the MARS, a 10-item scale assessing attitudes toward medication (e.g., It is unnatural for my mind and body to be controlled by medication.). The items scores were summed and averaged (range: 0-10). Scale: 0 (No) to 1 (Yes)
  Thompson K, Kulkarni J, Sergejew AA. Reliability and validity of a new Medication Adherence Rating Scale (MARS) for the psychoses. Schizophrenia Research. May 5 2000;42(3):241-247.
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: The number analyzed at each time point differs from the overall number enrolled due to participant drop out, clients who reported they are not prescribed medications for their mental health, and/or missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 170 | 213
  Baseline |  |  | 3.0 (1.7) | 3.3 (1.9)
  6 months: number analyzed (Participants) | 0 | 0 | 138 | 198
  6 months |  |  | 2.9 (1.9) | 3.2 (2.1)
  12 months: number analyzed (Participants) | 0 | 0 | 126 | 160
  12 months |  |  | 2.8 (1.7) | 3.1 (1.9)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.34, Mixed Models Analysis

24. Secondary Outcome: Health-Care Climate Questionnaire
Description: Perceived autonomy support was assessed with this 15-item scale (e.g., I am able to be open with [name] at our meetings.). Clients were prompted to report on the specific clinician from whose caseload they were randomly selected. The item scores were averaged. Scale: 1 (Strongly Disagree) to 7 (Strongly Agree)
  Williams GC, McGregor HA, King D, Nelson CC, Glasgow RE. Variation in perceived competence, glycemic control, and patient satisfaction: relationship to autonomy support from physicians. Patient Education & Counseling. Apr 2005;57(1):39-45.
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: The number analyzed at each time point differs from the overall number enrolled due to participant drop out and/or missing data. Some clients did not recall the clinician being asked about and/or discontinued treatment with that clinician during their study participation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 204 | 249
  Baseline |  |  | 6.0 (1.2) | 5.9 (1.1)
  6 months: number analyzed (Participants) | 0 | 0 | 155 | 200
  6 months |  |  | 5.8 (1.5) | 5.9 (1.2)
  12 months: number analyzed (Participants) | 0 | 0 | 82 | 130
  12 months |  |  | 6.0 (1.2) | 5.9 (1.3)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.71, Mixed Models Analysis

25. Secondary Outcome: Working Alliance Inventory (WAI)
Description: Perceived relatedness was assessed with this short form of the patient version of the WAI and is 12 items (e.g., We agree on what is important for me to work on.). Clients were prompted to report on the specific clinician from whose caseload they were randomly selected. The item scores were averaged. Scale: 1 (Never) to 7 (Always)
  Tracey TJ, Kokotovic AM. Factor structure of the Working Alliance Inventory. Psychological Assessment: A Journal of Consulting and Clinical Psychology. 1989;1(3):207.
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 202 | 248
  Baseline |  |  | 5.6 (1.2) | 5.5 (1.2)
  6 months: number analyzed (Participants) | 0 | 0 | 156 | 198
  6 months |  |  | 5.4 (1.4) | 5.6 (1.2)
  12 months: number analyzed (Participants) | 0 | 0 | 82 | 130
  12 months |  |  | 5.7 (1.3) | 5.6 (1.3)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.22, Mixed Models Analysis

26. Secondary Outcome: Working Alliance Inventory (WAI) - Tasks Subscale
Description: Perceived relatedness was assessed with this short form of the patient version of the WAI and has 12 items in total. This outcome is for the tasks subscale. Clients were prompted to report on the specific clinician from whose caseload they were randomly selected. The item scores were summed and averaged (range: 4-28). Scale: 1 (Never) to 7 (Always)
  Tracey TJ, Kokotovic AM. Factor structure of the Working Alliance Inventory. Psychological Assessment: A Journal of Consulting and Clinical Psychology. 1989;1(3):207.
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 202 | 248
  Baseline |  |  | 22.0 (5.4) | 21.5 (5.3)
  6 months: number analyzed (Participants) | 0 | 0 | 155 | 198
  6 months |  |  | 21.3 (6.4) | 22.2 (5.3)
  12 months: number analyzed (Participants) | 0 | 0 | 82 | 130
  12 months |  |  | 22.6 (5.6) | 22.4 (5.1)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.11, Mixed Models Analysis

27. Secondary Outcome: Working Alliance Inventory (WAI) - Goals Subscale
Description: Perceived relatedness was assessed with this short form of the patient version of the WAI and has 12 items in total. This outcome is for the goals subscale. Clients were prompted to report on the specific clinician from whose caseload they were randomly selected. The items scores were summed and averaged (range: 4-28). Scale: 1 (Never) to 7 (Always)
  Tracey TJ, Kokotovic AM. Factor structure of the Working Alliance Inventory. Psychological Assessment: A Journal of Consulting and Clinical Psychology. 1989;1(3):207.
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 201 | 246
  Baseline |  |  | 21.8 (5.1) | 21.4 (4.8)
  6 months: number analyzed (Participants) | 0 | 0 | 156 | 196
  6 months |  |  | 21.0 (5.4) | 21.8 (4.9)
  12 months: number analyzed (Participants) | 0 | 0 | 82 | 130
  12 months |  |  | 22.4 (5.0) | 21.7 (5.3)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.14, Mixed Models Analysis

28. Secondary Outcome: Working Alliance Inventory (WAI) - Bonds Subscale
Description: Perceived relatedness was assessed with this short form of the patient version of the WAI and has 12 items in total. This outcome is for the bonds subscale. Clients were prompted to report on the specific clinician from whose caseload they were randomly selected. The items scores were summed and averaged (range: 4-28). Scale: 1 (Never) to 7 (Always)
  Tracey TJ, Kokotovic AM. Factor structure of the Working Alliance Inventory. Psychological Assessment: A Journal of Consulting and Clinical Psychology. 1989;1(3):207.
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 203 | 247
  Baseline |  |  | 23.2 (5.1) | 23.0 (5.1)
  6 months: number analyzed (Participants) | 0 | 0 | 156 | 197
  6 months |  |  | 22.6 (6.5) | 23.0 (5.4)
  12 months: number analyzed (Participants) | 0 | 0 | 83 | 128
  12 months |  |  | 23.3 (5.5) | 22.8 (6.1)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.55, Mixed Models Analysis

29. Secondary Outcome: Patient Activation Measure-Mental Health (PAM-MH)-0 to 100 Scale
Description: Competence related to mental health management was assessed with the 13-item Patient Activation Measure-Mental Health (PAM-MH) (e.g., I know what each of my prescribed mental health medications does.). Each question was answered on a 4-point Likert-type scale: 1 (Strongly Disagree) to 4 (Strongly Agree). Higher scores=greater activation.
  Hibbard JH, Mahoney ER, Stockard J, Tusler M. Development and testing of a short form of the patient activation measure. Health Services Research. Dec 2005;40(6 Pt 1):1918-1930.
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 210 | 257
  Baseline |  |  | 62.5 (15.6) | 61.3 (14.8)
  6 months: number analyzed (Participants) | 0 | 0 | 184 | 230
  6 months |  |  | 63.6 (16.8) | 62.1 (17.3)
  12 months: number analyzed (Participants) | 0 | 0 | 164 | 206
  12 months |  |  | 64.8 (15.4) | 65.2 (16.9)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.91, Mixed Models Analysis

30. Secondary Outcome: Short-Form Health Survey (SF-12)-Physical Health Functioning
Description: Physical and mental health functioning was assessed with the Short Form 12-Item Health Survey (SF-12). The SF-12 is a health-related quality of life measure, derived from the 36-item Medical Outcomes Study survey and containing items yielding a Mental Health Component Score and a Physical Health Component Score. Higher composite scores indicate higher health-related quality of life. Items are weighted and then transformed into norm-based scores (range: 0-100).
  Ware JE, Jr. , Kosinski M, Keller SD. A 12-item short-form health survey: Construction of scales and preliminary tests of reliability and validity. Medical Care. 1996;34(3):220 -233.
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline |  |  | 41.4 (8.7) | 41.9 (7.9)
  6 months: number analyzed (Participants) | 0 | 0 | 186 | 234
  6 months |  |  | 42.3 (8.3) | 41.8 (7.8)
  12 months: number analyzed (Participants) | 0 | 0 | 168 | 209
  12 months |  |  | 42.0 (7.9) | 41.7 (7.8)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.48, Mixed Models Analysis

31. Secondary Outcome: Short-Form Health Survey (SF-12)-Mental Health Functioning
Description: as for outcome 30
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline |  |  | 42.6 (7.8) | 42.0 (8.1)
  6 months: number analyzed (Participants) | 0 | 0 | 186 | 234
  6 months |  |  | 42.7 (7.7) | 43.0 (8.0)
  12 months: number analyzed (Participants) | 0 | 0 | 168 | 209
  12 months |  |  | 43.2 (7.2) | 43.4 (8.0)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.67, Mixed Models Analysis

32. Secondary Outcome: Patient Health Questionnaire 9-item (PHQ-9)
Description: The PHQ-9 is a brief, self-report assessment. It provides a summed total score that indicates likelihood of major depressive disorder. Scores ≥10 are considered a positive screen (sensitivity 88%, specificity 88%) and also effectively measures response to treatment (<5 indicate remission, of 5-9 indicate partial response, and ≥10 indicates no response). Item scores are summed and averaged (range: 0-27). Scale: 0 (Not at all), 1 (Several days), 2 (More than half the days), 4 (Nearly every day). When problems are identified, the difficulty of those problems are rated on 4 point scale (Not difficult at all to Extremely difficult).
  Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. Journal of General Internal Medicine. Sep 2001;16(9):606-613.
  American Psychiatric Association. Diagnostic and statistical manual of mental disorders - Text Revision (4th ed.). Washington, DC: American Psychiatric Association; 2000.
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 197 | 238
  Baseline |  |  | 9.6 (5.9) | 10.0 (6.0)
  6 months: number analyzed (Participants) | 0 | 0 | 165 | 197
  6 months |  |  | 8.8 (6.1) | 9.8 (6.3)
  12 months: number analyzed (Participants) | 0 | 0 | 146 | 183
  12 months |  |  | 9.1 (6.0) | 9.4 (5.8)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.77, Mixed Models Analysis

33. Secondary Outcome: Generalized Anxiety Disorder (GAD-7)
Description: Anxiety was assessed with the 7-item Generalized Anxiety Disorder (GAD-7). It can be scored continuously on a 0-21 severity scale and cutpoints have been established for estimating the probability of the 4 most common and clinically relevant anxiety disorders - generalized anxiety disorder, panic disorder, post-traumatic stress disorder, and social anxiety disorder. Scale: 0 (not at all), 1 (several days), 2 (more than half the days), 3 (nearly every day)
  Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Archives of Internal Medicine. May 22 2006;166(10):1092-1097.
  Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. Mar 6 2007;146(5):317-325.
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 181 | 216
  Baseline |  |  | 9.4 (5.7) | 9.7 (5.9)
  6 months: number analyzed (Participants) | 0 | 0 | 145 | 194
  6 months |  |  | 8.5 (5.7) | 8.4 (5.6)
  12 months: number analyzed (Participants) | 0 | 0 | 147 | 173
  12 months |  |  | 8.5 (5.8) | 8.8 (5.5)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.59, Mixed Models Analysis

34. Secondary Outcome: Client Satisfaction Questionnaire
Description: Engagement was assessed with patient satisfaction using the Client Satisfaction Questionnaire, an 8-item satisfaction checklist (e.g., How would you rate the quality of service you have received? and, If a friend were in need of similar help, would you recommend [name of agency] to him or her?). The item scores were averaged. Scale: 1 to 4 with response text dependent upon the question (e.g., 1-Poor to 4-Excellent, 1-No, definitely not to 4-Yes, definitely, or 1-Quite dissatisfied to 4-Very satisfied).
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 211 | 257
  Baseline |  |  | 3.4 (0.6) | 3.5 (0.5)
  6 months: number analyzed (Participants) | 0 | 0 | 177 | 225
  6 months |  |  | 3.4 (0.6) | 3.5 (0.5)
  12 months: number analyzed (Participants) | 0 | 0 | 168 | 208
  12 months |  |  | 3.5 (0.5) | 3.5 (0.5)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.64, Mixed Models Analysis

35. Secondary Outcome: Quality of Care-Person Centered Care
Description: Perceived Quality of Care was assessed with a 31 item scale (e.g., Staff spent extra time with me when I needed them.). This scale for clients was adapted from the one developed for staff. Person Centered Care was measured with a subset of questions from this scale. The item scores were averaged. Scale: 0 (never) to 5 (always)
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 210 | 255
  Baseline |  |  | 3.8 (1.1) | 3.8 (1.0)
  6 months: number analyzed (Participants) | 0 | 0 | 185 | 232
  6 months |  |  | 3.7 (1.1) | 3.8 (1.1)
  12 months: number analyzed (Participants) | 0 | 0 | 161 | 202
  12 months |  |  | 3.6 (1.1) | 3.9 (1.1)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.05, Mixed Models Analysis

36. Secondary Outcome: Quality of Care-Negative Interactions
Description: Perceived Quality of Care was assessed with a 31 item scale (e.g., Staff spent extra time with me when I needed them.). This scale for clients was adapted from the one developed for staff. Negative Interactions were measured with a subset of questions from this scale. Item scores were averaged. Scale: 0 (never) to 5 (always)
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 209 | 257
  Baseline |  |  | 4.3 (0.9) | 4.3 (0.8)
  6 months: number analyzed (Participants) | 0 | 0 | 185 | 232
  6 months |  |  | 4.8 (0.8) | 4.3 (0.9)
  12 months: number analyzed (Participants) | 0 | 0 | 160 | 202
  12 months |  |  | 4.3 (0.8) | 4.4 (0.9)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.06, Mixed Models Analysis

37. Secondary Outcome: Quality of Care-Inattentive Care
Description: Perceived Quality of Care was assessed with a 31 item scale (e.g., Staff spent extra time with me when I needed them.). This scale for clients was adapted from the one developed for staff. Inattentive care was measured with a subset of questions from this scale. Item scores were averaged. Scale: 0 (never) to 5 (always)
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 210 | 258
  Baseline |  |  | 4.2 (0.9) | 4.2 (0.8)
  6 months: number analyzed (Participants) | 0 | 0 | 183 | 233
  6 months |  |  | 4.3 (0.7) | 4.3 (0.8)
  12 months: number analyzed (Participants) | 0 | 0 | 161 | 200
  12 months |  |  | 4.2 (0.8) | 4.3 (0.8)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.84, Mixed Models Analysis

38. Secondary Outcome: Quality of Care Total
Description: Perceived Quality of Care was assessed with a 31 item scale (e.g., Staff spent extra time with me when I needed them.) and then refined to 22 items through data collected and analyzed in this study. This scale for clients was adapted from the one developed for staff. Item scores were averaged. Scale: 0 (never) to 5 (always)
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
units on a scale
  Baseline: number analyzed (Participants) | 0 | 0 | 209 | 257
  Baseline |  |  | 4.0 (0.8) | 4.0 (0.8)
  6 months: number analyzed (Participants) | 0 | 0 | 185 | 233
  6 months |  |  | 4.0 (0.8) | 4.0 (0.8)
  12 months: number analyzed (Participants) | 0 | 0 | 161 | 202
  12 months |  |  | 3.9 (0.9) | 4.1 (0.8)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.14, Mixed Models Analysis

39. Secondary Outcome: Patient Engagement-Missed Appointments
Description: Patient engagement was assessed by the proportion of missed appointments (when the client cancelled or did not show for a scheduled appointment divided by the total scheduled). This data was retrieved from client medical records at the agencies. Data from 3 time periods were analyzed (6 months prior to baseline through baseline, baseline to 6 months, and 6 months to 12 months). The below table illustrates the missed appointments for each time period.
Time Frame: Measured with clients at baseline, 6 months, and 12 months
Population: The number analyzed at each time point differs from the overall number enrolled due to missing data (medical records not available) and clients discontinuing treatment at their respective agency.
Measure: Mean (Standard Deviation); unit: appointments at mental health agency
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
Number analyzed (Participants) | 0 | 0 | 211 | 258
appointments at mental health agency
  Baseline: number analyzed (Participants) | 0 | 0 | 203 | 250
  Baseline |  |  | 11.96 (12.51) | 11.02 (12.68)
  6 months: number analyzed (Participants) | 0 | 0 | 202 | 247
  6 months |  |  | 14.47 (15.93) | 12.20 (14.91)
  12 months: number analyzed (Participants) | 0 | 0 | 185 | 233
  12 months |  |  | 14.52 (15.85) | 11.50 (16.08)
Statistical Analysis 1: Comparison: BREATHE-Clients vs Motivational Interviewing-Clients; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.45, Mixed Models Analysis

ADVERSE EVENTS:
Description: Adverse events were not monitored or assessed for any participants in this minimal risk study. However, we did become aware of clients who had died during the study during data collection periods for follow-up interviews. The deaths were not related to the study.
Groups:
- BREATHE-Mental Health Care Staff: Mental Health Care Staff randomized to the BREATHE intervention Staff were invited to attend an 8-9 hour BREATHE workshop delivered in 3 sessions, each about one month apart. Staff were asked to complete online surveys at the following time points: Baseline, 3 months, 6 months, and 12 months.
- BREATHE-Clients: Clients linked to staff randomized to the BREATHE intervention Clients were invited to be interviewed at the following time points: Baseline, 6 months, and 12 months.
- Motivational Interviewing-Clients: Clients linked to staff randomized to the MI intervention Clients were invited to be interviewed at the following time points: Baseline, 6 months, and 12 months.
Arm/Group | BREATHE-Mental Health Care Staff | Motivational Interviewing-Mental Health Care Staff | BREATHE-Clients | Motivational Interviewing-Clients
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/103 | 4/211 | 4/258
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Absence of treatment as usual condition, high staff turnover, and difficulty linking patients with specific clinicians with whom they had meaningful contact

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes